CLINICAL TRIAL: NCT03885609
Title: Safety and Efficacy of the ToothWave Power Toothbrush for Extrinsic Stain Reduction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Home Skinovations Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DO116028A
Record Dates: First submitted 2019-03-20; First posted 2019-03-21 (Actual); Last update posted 2019-09-10 (Actual); Status verified 2019-03

CONDITIONS: Tooth Discoloration
MeSH Terms: conditions — Tooth Discoloration

STUDY DESIGN:
Intervention Model Description: Double arm, single blind prospective study
Who Masked: Outcomes Assessor
Masking Description: The Outcomes Assessors will not be exposed to the type of brush the subject is using or to the group they are assigned to (treatment or control).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment - toothwave brush (Experimental): Subjects using the Silk'n ToothWave RF utilizing toothbrush
  Interventions: Device: ToothWave
- Control - powered toothbrush (Sham Comparator): Subject using a regular powered toothbrush with no RF.
  Interventions: Device: powered toothbrush

INTERVENTIONS:
Device: ToothWave — RF-utilizing powered toothbrush for teeth whitening
  Other Names: RF toothbrush
  Arms: Treatment - toothwave brush
Device: powered toothbrush — regular powered toothbrush with no RF
  Arms: Control - powered toothbrush

SUMMARY:
This study is a single blind, prospective study aimed to evaluate the safety and efficacy of the Silk'n ToothWave Power Toothbrush for stains reduction and improvement of teeth shade.

DETAILED DESCRIPTION:
The study includes 84 treatment sessions, twice a day, and 4 clinic visits over a period of 6 weeks.

One treatment group (Silk'n power toothbrush - ToothWave) and 1 control group (an ADA approved power toothbrush (PTB)) will participate in the study.

For each patient, efficacy assessment data will be collected at baseline, 4 weeks, and at 6 weeks. The average stain data will be calculated for each group.

Treatment is defined as a timed, 2 minute brushing of the teeth according to the manufactur-er's instructions, twice daily (morning and evening). Brushing will be undertaken using the Silk'n toothbrush and standard fluoride toothpaste. The control group will use an ADA ac-cepted PTB and the same standard fluoride toothpaste.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects aged 18-70, that are in good health.
2. Subjects should have notable extrinsic dental stains on the front teeth with a total extrin-sic facial tooth stain score ≥14 according to the LSI.
3. The subjects should understand the information provided about the investigative nature of the treatment, possible benefits and side effects. Subjects will sign the Informed Consent Form.
4. The subjects should be willing to comply with the study procedure and schedule, includ-ing the follow up visits, and will refrain from using any other teeth whitening technologies during this period.
5. The subject did not perform any procedure for teeth whitening (either at home or in clin-ic) at least 3 years prior to participating in the study

Exclusion Criteria:

1. Any condition that might make it unsafe for the subject to participate in the study, at the discretion of the investigator
2. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
3. Pregnant or nursing by subject report.
4. Any active condition in the oral cavity at the discretion of the investigator.
5. Any surgery in the treated area within 3 months prior to treatment, or before complete healing.
6. Subjects that do not brush regularly.
7. Regular tobacco smokers.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-02-28 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Extrinsic Stains | 6 weeks
  Extrinsic Stains will be evaluated using the validated Lobene Stain Index (LSI)
  Stain Intensity score range is between 0 and 3, where:
  0 = no stain
  1. = light stain
  2. = moderate stain
  3. = heavy stain
  The mean stain intensity will be calculated for both the gingival and body regions of the incisor teeth for each subject.
  Stain Area score rage is between 0 and 3, where:
  0 = no stain
  1. = stain covering up to one third of region
  2. = stain covering up to two thirds of region
  3. = stain covering more than two thirds of region
  The mean stain area will be calculated for both the gingival and body regions of the incisor teeth for each subject.

SECONDARY OUTCOMES:
Tooth color assessment | 6 weeks
  VITA Bleachedguide 3D-Master shade guide, includes 29 shade levels defined by the American Dental Association (ADA). These shade levels represents the brightness of the tooth where 1 is the whitest and 29 is the darkest shade.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffery L Milleman, DDS, MPA, Principal Investigator — Salus research center
Locations (1):
- Salus research, Fort Wayne, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Amaechi BT, Levi L, Silman Z, Evans V, Shehata MAS, Alonso-Ryan JR, Phillips TS, Ugwokaegbe PC, Farokhi MR. Clinical efficacy of a novel radiofrequency toothbrush for tooth stain reduction and tooth whitening: A randomized controlled trial. J Am Dent Assoc. 2022 Apr;153(4):342-353. doi: 10.1016/j.adaj.2021.09.006. Epub 2021 Dec 29. PMID 34973707